CLINICAL TRIAL: NCT06826183
Title: The Use of Activity and Impedance From a Continuous, Implantable Sensor to Detect Deterioration in Asymptomatic Patients With Severe Aortic Stenosis (AS) Under a Watchful Waiting Program
Brief Title: Implantable Sensor in Aortic Stenosis
Acronym: ISAS
Status: Completed | Type: Observational
Sponsor: Barts & The London NHS Trust (Other)
Collaborators: East Sussex Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 011760
Record Dates: First submitted 2019-01-23; First posted 2025-02-13 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Aortic Stenosis
Keywords: cardiopulmonary exercise testing; biomarker
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: REVEAL Linq device — Implantable loop recorder

SUMMARY:
To establish the relationship between a panel of biological markers obtained from the REVEAL Linq device and exercise performance as judged by cardiopulmonary exercise testing

DETAILED DESCRIPTION:
Patients with severe aortic stenosis (AS) and symptoms have a poor prognosis without surgical or percutaneous intervention; however patients with severe asymptomatic aortic stenosis can be managed conservatively until the severity worsens to a critical extent. Following these patients up is challenging and inexact, and many methods have been proposed to predict an early deterioration. These include exercise testing, the demonstration of a significant increase in mean gradient across the valve on exercise and biomarkers such as Brain Natriuretic peptide (BNP). Current guidelines suggest that aortic valve surgery should be performed on the basis of symptoms in patients with severe aortic stenosis and even in the absence of symptoms in those with very severe disease. The use of treadmill exercise testing is also advocated to establish the presence of unrecognised symptomatic limitation (Class IIa). The complexity of this process, and the risks posed by severe aortic stenosis with symptoms, lead some authorities recommending surgery on all patients with severe aortic stenosis regardless of symptoms in the presence of evidence of rapid progression.

The burden of aortic stenosis is high in developed countries and increasing because of improved survival and greater longevity. As the population ages the prevalence of disease will become highly significant as moderate or severe AS can be demonstrated in 7% of patients over the age of 75 years, and severe aortic valve (AV) calcification seen in 17-19% of the over 80s. The follow up of these patients is often labour intensive, and variably performed. Consensus statements from the British Heart Valve Society and the European Working Party on Valvular Heart Disease recommend follow up in specialist valve clinics, but contemporary UK data suggest that these are few and far between .

There remains a significant group of patients who die or deteriorate while waiting for interventions and the overall mortality is higher in AS patients than in other forms of heart valve disease. The cause for mortality in patients with AS is believed to be haemodynamic collapse, however a higher rate of symptomless arrhythmic events has been noted in this population including bradyarrhythmias, atrial fibrillation and ventricular arrhythmias; the total burden being around 17% in TAVI candidates on a single 24 Holter monitor. This is unsurprising as part of the pathological process underlying AS includes fibrosis of the left ventricular and especially the septal myocardium.

The principle methods of assessment for patients with severe aortic stenosis remain a resting echocardiogram and clinical assessment. Asymptomatic patients may also be assessed with an exercise treadmill test. However, there is concern that asymptomatic patients may deteriorate or have events between follow up visits, or that adequate follow up arrangements may be difficult to achieve.

Continuous or implantable biological measurement and monitoring is a well-established concept and has been available on pacing devices and used in routine clinical practice for some years. The factor that has limited the usefulness of automatic detection algorithms for identifying deterioration in heart failure remains the large variability in clinical status from day to day, such that a true deterioration may become lost amongst a large number of minor clinical insignificant daily fluctuations. In aortic stenosis however, the situation is different. The disease has an inexorable progression and the presence of symptoms defines the need for definitive therapy. This therefore presents a different objective for device monitoring which is required to demonstrate clear evidence of progressive deterioration in order to justify definitive therapy, rather than the day to day optimisation of heart failure medication.

Many measurable parameters are associated with deterioration in patients with heart failure including increasing heart rate, deteriorating autonomic function and reduced daily activity. The use of these continuous monitored biological variables both available on the REVEAL and Linq devices can be integrated into a multiparameteric model to describe the clinical deterioration in aortic stenosis. This, coupled to a better description of the presence of arrhythmic events, provides an exciting new opportunity, if validated, to improve the care of these patients and aid clinical decision making during longitudinal follow up.

ELIGIBILITY:
Inclusion Criteria:

1. Severe aortic stenosis defined as effective orifice area (EOA) < 1.0 cm2 (or 0.6 cm2/m2 when indexed for body surface area) and peak velocity > 4.0 m/s or mean gradient > 40mmHg
2. No AS attributable symptoms during clinical consultation
3. Informed consent
4. Aged 18 years of age or over

Exclusion Criteria:

1. Left ventricular ejection fraction <50%
2. Severe mitral regurgitation
3. PA systolic pressure >40mmHg
4. Ischaemic heart disease with evidence of ongoing ischaemia
5. Anginal chest pain
6. Inability to cycle
7. Unrecordable echo windows
8. Alternative pathology like to be life limiting within 2 years
9. Chronic renal failure (EGFR<30)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Asymptomatic severe aortic stenosis
Sampling Method: Non-Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2017-08-15 (Actual); Primary Completion 2019-03-09 (Actual); Study Completion 2020-03-09 (Actual)

PRIMARY OUTCOMES:
To establish the relationship between a panel of biological markers obtained from the REVEAL Linq device and exercise performance as judged by cardiopulmonary exercise testing. | 12 months
The regressive relationship between total weekly activity from the Reveal Linq and change in VO2 peak /Oxygen Uptake Efficiency Slope (OUES) established by cardiopulmonary exercise testing between visits. | 12 months

SECONDARY OUTCOMES:
The relationship between weekly heart rate variability and VO2 peak /OUES | 12 months
The relationship between weekly heart rate and VO2 peak /OUES | 12 months
The relationship between acoustic murmur intensity and VO2 peak /OUES | 12 months
The relationship between S1/S2 intensity and VO2 peak/ OUES | 12 months
The relationship between murmur intensity augmentation and VO2 peak/OUES | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Guy Lloyd, Principal Investigator — Barts & The London NHS Trust
Locations (1):
- Barts Health NHS Trust, London, United Kingdom